CLINICAL TRIAL: NCT07050797
Title: Using Data-driven Insights From Wearable Technologies to Inform Whole School Physical Activity Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other); University of Bristol (Other); Loughborough University (Other)
Responsible Party: Principal Investigator, Georgina Wort, Doctoral Researcher, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EP 22 018
Record Dates: First submitted 2022-10-07; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Physical Inactivity
Keywords: Mixed-methods; Whole-school; Wearable Technology; Co-design
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The first two-weeks within each school children's baseline physical activity data will be collected. Children and school staff will be blinded to the data, receiving no feedback. Teachers will be instructed not to change normal school practices or encourage children's physical activity.
  In control groups pupils will continue to wear the monitors for another 3-weeks, with children and school staff continuing to be blinded to the data.
- Whole-School Intervention (Experimental): After the 2-week baseline, schools will be assigned to either control or intervention groups. For schools in the intervention group pupils' baseline physical activity data will be shared with staff during focus groups and strategies which aim to improve pupils' physical activity will be co-designed with the PI. These individualised whole-school strategies will then be implemented over the subsequent 3-weeks. During this time staff will be able to access pupils' physical activity data through the accompanying software application, which will be installed on school computers, with the ability to continue refining strategies.
  Interventions: Behavioral: Individualised whole-school intervention, developed using data sharing and co-design.

INTERVENTIONS:
Behavioral: Individualised whole-school intervention, developed using data sharing and co-design. — Individualised whole-school intervention, developed using data sharing and co-design.
  Arms: Whole-School Intervention

SUMMARY:
This is a whole-school study using co-design to inform tailored school-based interventions. Schools will be allocated either to a control or intervention group and KS2 pupils will be asked to wear a wrist-worn physical activity monitor for a total of 5-weeks. During this time the PI will be present in schools to collect notes regarding school practices and daily variation. In the control groups pupils will wear monitors for 5-weeks (blinded to data) and school practice will continue as normal; school staff will be asked not to make any changes within school. After these 5-weeks, schools' will receive a detailed report about pupils' physical activity, and a researcher will come in to discuss findings. In the intervention groups pupils will wear monitors for 2-weeks (blinded to data). After this time the PI will present staff with pupils' physical activity during a focus group in the form of user-friendly graphs and a summary report. Staff will be asked to reflect on school practices and co-design feasible and practical strategies to improve pupils' physical activity. These strategies will then be implemented over the following 3-weeks, with immediate physical activity feedback on the accompanying software application, which will be installed on school computers, and support from the PI. At the end of the 5th week, during another focus group, schools will be given a summary of the data and changes in pupils' physical activity. This is where staff can reflect on the project and highlight challenges or barriers, and strategies they believed to be successful. The researcher will not prescribe any changes, this will be at the initiation of the school and staff members.

DETAILED DESCRIPTION:
This is a whole-school study which will follow a randomised controlled design and use co-design to inform tailored school-based interventions. Stratified randomisation will be used to allocate each school to either control or intervention groups. Interventions will be co-designed during focus groups in which pupils' baseline physical activity data will be discussed with their school staff members.

After the first two schools have been randomly assigned, minimisation will be used to allocate schools to either intervention or control groups. Minimising aims at specifically minimising differences in group variates. After the first two schools have been randomly allocated, it will be determined whether the subsequent allocation of schools would lead to a better balance in the variables of interest between control and intervention groups. For this study the variables of interest will be the school size (grouped into small, medium, and large) and free school meal (used as a marker of deprivation and grouped into low, medium, or high). The imbalance of these variables between control and intervention groups will be minimised by allocating schools to the group with the smaller total of the relevant variable (or at random if the totals are the same). When initially recruiting, schools will be informed about the possibility of being assigned to either the control or intervention group. Consent forms will be obtained from staff and parents/carers before the school is assigned to control or intervention.

All schools involved in the project will complete 2-weeks of baseline physical activity measures. During this time pupils involved in the project will wear Moki Technology physical activity bands within school hours only. Pupils and teachers will be blinded to the physical activity data, receiving no feedback or insights into how active they are. During this time the lead researcher will also fill out a diary each week with the help of teachers and staff members to detail what happens each school day and other factors, including weather. The purpose of this is so that when presented with the physical activity data members of staff can recall more easily what happened within the school day to explain any physical activity differences. Using a diary is not intended to prompt staff members to reflect on, or change physical activity within the school day, therefore, staff members will be told this is to detail all the commitments within the school day and to understand normal school practices.

Observational methods/ ethnographic style research will also be carried out during this time by the lead researcher to gain a greater insight into school practices and physical activity opportunities. The notes collected will be used to inform the later focus group and co-design of strategies.

Control Group: Those involved in the control group will continue to wear the bands for another 3-weeks following the baseline measures, receiving no feedback on their physical activity. Following this 5-week period in total, control groups will get a detailed overview of their pupils' physical activity in the form of user-friendly, visually appealing graphs, alongside personalised suggestions for improving physical activity metrics, and the opportunity to discuss results with the researcher if they wish. This is so they also get value from the project and can use the data to inform their future school practices. However, for the purpose of this study, no changes will be made to school practices for the duration they are involved with the project. Control schools will be told not to make any changes to policy or practices; it will be explained that we are trying to get an accurate representation of schools' physical activity, rather than making any changes at this stage.

Intervention Group: Staff members in intervention schools will be involved in focus groups where pupils' physical activity data from baseline measures and a reference data set will be shared, and an intervention co-designed during the focus groups conducted after the 2-week baseline measures. The focus groups will be conducted with teachers, leadership, and wider staff and lead by the researcher. A member of staff (i.e., P.E. lead) will be asked to act as school lead for the project, their role to ensure the research design and intervention are followed. They will be asked about their views of children's physical activity and school's influence before getting their views on the physical activity data, what they think are the barriers and facilitators to physical activity within their school, and what they think could be done to help encourage activity and address inequalities. The Creating Active School Framework (Daly-Smith et al., 2020) will be used during focus groups to help individuals think of aspects of the school day which could be adapted to improve pupils' physical activity outcomes. At the end of this focus group an intervention, which is co-designed, and contains at least 3 strategies which map onto the creating active schools' framework, will be implemented in the following 3-weeks.

During the 3-weeks intervention phase, the school staff will have access to the live physical activity data returned from the activity bands through the accompanying software application (which will be installed on their computers). This will be to enable self-monitoring by feeding back physical activity data. During the first week the researcher will support the schools in how to use the software, understand the data, and will provide guidance on how it could be used to further develop their practices at both school and class level.

Observational/ ethnographic methods will be conducted throughout the 5-week duration in both control and intervention schools to gain an understanding of school practices, the opportunities for children's physical activity and to ensure either normal school practices are being maintained or to assess intervention fidelity. Handwritten notes will be taken, before more detailed notes are subsequently typed up; no personal or sensitive information will be collected.

Daly-Smith A, Quarmby T, Archbold VS, Corrigan N, Wilson D, Resaland GK, et al. Using a multi-stakeholder experience-based design process to co-develop the Creating Active Schools Framework. Int J Behav Nutr Phy. 2020;17(1):13.

ELIGIBILITY:
Inclusion Criteria:

* Any KS2 pupil from the UK schools recruited.

Exclusion Criteria:

* No exclusion criteria.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 549 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Changes-1 | change between baseline (assessed for 3-weeks) and during intervention period (assessed for 3-weeks) within each school
  Daily step counts

SECONDARY OUTCOMES:
Qualitive Data | following baseline and intervention measures (~1-2hr focus group workshop)
  During focus groups teachers and staff will be asked for their responses to physical activity data, what strategies they believe would be feasible and acceptable to implement within their school environment, what challenges, barriers were faced when implementing and which strategies they perceived as successful.
Physical Activity Changes-2 | changes from baseline (assessed for 3-weeks) and during intervention period (assessed for 3-weeks) within each school
  Moderate to Vigorous Physical Activity (MVPA) minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF